CLINICAL TRIAL: NCT06095440
Title: A Retrospective Analysis of Outcomes in Patients with Hepatorenal Syndrome At Methodist Dallas Medical Center
Status: Recruiting | Type: Observational
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 020.HEP.2023.D
Record Dates: First submitted 2023-07-06; First posted 2023-10-23 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-08

CONDITIONS: Hepatorenal Syndrome
MeSH Terms: conditions — Hepatorenal Syndrome | interventions — Liver Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Hepatorenal Syndrome outcome in Patients at Methodist Health systems — 1.2.1. To perform a retrospective analysis of patients with HRS with the aim of comparing various treatment modalities such as vasoconstrictors, albumin, CRRT, Molecular Adsorbent Recirculating System (MARS), and TIPS.
  Other Names: liver transplantation

SUMMARY:
Hepatorenal syndrome (HRS) is a common cause of acute kidney injury (AKI) in patients with liver disease [1]. Increased activity and presence of vasodilators such as nitric oxide in cirrhotic patients leads to vasodilation, especially in the splanchnic circulation, resulting in hemodynamic changes that precipitate renal injury [1]. Patients may present with elevated serum creatinine (Cr), benign urine sediment, and low urine sodium [1].

DETAILED DESCRIPTION:
There are two main classifications of HRS: HRS-AKI (previously known as type 1 HRS) and diuretic-resistant ascites (previously known as type 2 HRS) [1].

The ultimate treatment for patients with HRS is to improve hepatic function via treatment of underlying etiology or liver transplantation; however, this is not always immediately possible due to the high demand for liver transplantation among other factors [1]. Continuous renal replacement therapy (CRRT) can also be considered, especially in patients with severe electrolyte derangements such as hypokalemia or pulmonary edema, that are not responding to medical therapy [1]. Often, CRRT is used as a bridging therapy to stabilize patients until they are optimized for receiving a liver transplant [1, 2]. CRRT, however, comes with its own risks and disadvantages such as hypotension and increased risk of cardiac adverse events [2]. In certain cases, transjugular intrahepatic portosystemic shunts (TIPS) can benefit patients with HRS by reducing portal pressure resulting in increase in renal perfusion [1].

ELIGIBILITY:
Inclusion Criteria:

* All patients >18 years old that were hospitalized between April 1st 2019 and April 1st 2023 who either presented with HRS-AKI or developed a diagnosis of HRS during the hospital course. HRS-AKI will be defined based on the ICA criteria, described below:

  1. Presence of cirrhosis, acute liver failure, or acute-on-chronic liver failure
  2. An increase in serum Cr of ≥0.3 mg/dL within 48 hours or ≥50% from baseline value and/or urinary output ≤0.5 mL/kg of body weight for ≥6 hours (requires use of a urinary catheter)
  3. No full or partial response for ≥2 days of diuretic withdrawal and volume expansion with albumin (dosed at 1 g/kg of body weight/day)
  4. Absence of shock
  5. No current or recent treatment with nephrotoxic drugs
  6. Absence of parenchymal renal disease
  7. Suggestion of renal vasoconstriction based on FENa <0.2%

Exclusion Criteria:

* 1. HRS-AKI patients <18 years of age 2. All patients hospitalized between April 1st 2019 and April 1st 2023 without a diagnosis of HRS-AKI.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: - All patients >18 years old that were hospitalized between April 1st 2019 and April 1st 2023 who either presented with HRS-AKI or developed a diagnosis of HRS during the hospital course. HRS-AKI will be defined based on the ICA criteria, described below:
  1. Presence of cirrhosis, acute liver failure, or acute-on-chronic liver failure
  2. An increase in serum Cr of ≥0.3 mg/dL within 48 hours or ≥50% from baseline value and/or urinary output ≤0.5 mL/kg of body weight for ≥6 hours (requires use of a urinary catheter)
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-05-13 (Actual); Primary Completion 2025-05-13 (Estimated); Study Completion 2025-05-13 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome for HRS-AKI patients | 4 years
  Mortality rates, morbidities, complications, and other clinically relevant outcomes in HRS-AKI patients

SECONDARY OUTCOMES:
post transplant mortality rates | 4 years
  post-transplant mortality rates HRS-AKI-associated costs

CONTACTS AND LOCATIONS:
Overall Officials: Parvez Mantry, MD, Principal Investigator — Methodist Health System
Locations (1):
- Liver Institute of Methodist Dallas Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No